CLINICAL TRIAL: NCT07023965
Title: Multicenter Cohort Long-term Follow-up Study of Participants From Phase III Clinical Trials of Donaperminogene Seltoplasmid Injection for Critical Limb Ischemia
Brief Title: Follow-up Study Using Gene Therapy for Critical Limb Ischemia (NL003-CLI-III-L)
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NL003-CLI-III-L
Record Dates: First submitted 2025-06-06; First posted 2025-06-17 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Arterial Disease(PAD); Arterial Occlusive Disease; Arteriosclerosis Obliterans; Thromboangiitis Obliterans; Diabetic Foot Ulcer (DFU); Diabetic Foot Ulcer Ischemic; Critical Limb Ischemia (CLI)
Keywords: HGF; Critical Limb Ischemia; Gene therapy
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases; Arteriosclerosis Obliterans; Thromboangiitis Obliterans; Diabetic Foot; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants exposed to drug NL003 from Phase III Clinical Trials
  Interventions: Drug: NL003
- Participants exposed to placebo from Phase III Clinical Trials
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NL003 — This is an observational study, and the interventions have already been administered in the preceding Phase III clinical trials.
  Groups: Participants exposed to drug NL003 from Phase III Clinical Trials
Drug: Placebo — This is an observational study, and the interventions have already been administered in the preceding Phase III clinical trials.
  Groups: Participants exposed to placebo from Phase III Clinical Trials

SUMMARY:
The goal of this observational study is to learn about the long-term effects of Donaperminogene Seltoplasmid Injection (NL003) in participants who have been received drug NL003 or placebo at least one dose from the parent phase III clinical study to treat their critical limb ischemia (CLI). The main questions it aims to answer are:

* First, what medical problems do participants have after taking drug NL003 to treat CLI?
* Second, does drug NL003 make CLI participants live longer without serious problems (amputations or target vessel revascularizations) ?

Participants who have already received drug NL003 for CLI will complete online surveys about their health conditions. This study will continue until at least 36 months after the participant's first dose.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, long-term follow-up cohort study. A remote follow-up system is recommended as a tool for the study, however, in-person visits or phone calls at the research center will be conducted if remote follow-up is not feasible. The study will retrospectively collect data from the last visit in the parent Phase III study and prospectively gather data following informed consent. It will continue until at least 36 months after the first dose administered to the last enrolled participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have previously enrolled in Phase III clinical trials of recombinant human hepatocyte growth factor plasmid injection (Donaperminogene Seltoplasmid Injection) for the treatment of critical limb ischemia (including ulcers and rest pain) and have received at least one dose of the treatment.

Exclusion Criteria:

* Participants who refused to provide written informed consent;
* Participants who refused to cooperate with the retrospective or prospective data collection.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were enrolled from the parent phase III clinical study identified by protocol numbers NCT04274049 and NCT04275323.
Sampling Method: Non-Probability Sample
Enrollment: 542 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Incidence of benign and malignant tumors | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Incidence of significant vision loss, blindness, or other obvious visual abnormalities | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Incidence of major cardiovascular and cerebrovascular events | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Pregnancy status and its outcomes | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Amputation-free survival of the trial limb | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
  Amputation-free survival of the trial limb is one of the key endpoints for efficacy assessment. The time from the first dose administration to the occurrence of amputation above the ankle of the trial limb or death due to any cause, whichever occurs first.
Amputation-free survival or target vessel revascularization composite endpoint | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
  Amputation-free survival or target vessel revascularization composite endpoint is one of the key endpoints for efficacy assessment. The time from the first dose administration to the occurrence of amputation above the ankle of the trial limb, death due to any cause, or target vessel revascularization* of the trial limb, whichever occurs first.*Target vessel revascularization: bypass grafting, endovascular revascularization, thrombectomy, or thrombolysis of the trial limb.
Amputation-free survival or target vessel revascularization or neovascularization therapies (including stem cell or gene therapy) composite endpoint | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
  Amputation-free survival or target vessel revascularization or neovascularization therapies (including stem cell or gene therapy) composite endpoint is one of the key endpoints for efficacy assessment. The time from the first dose administration to the occurrence of amputation above the ankle of the trial limb, death due to any cause, or target vessel revascularization and neovascularization therapies (including stem cell or gene therapy) of the trial limb, whichever occurs first.

SECONDARY OUTCOMES:
All-cause mortality rate, time to death | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Major amputation rate of the trial limb (amputation plane above the ankle) | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Minor amputation rate of the trial limb (below the ankle, including toe amputation) | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Incidence of target vessel revascularization of the trial limb | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Rehospitalization rate for worsening ischemic symptoms of the trial limb | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Incidence of death due to acute myocardial infarction or stroke | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Time to amputation of the trial limb | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Level of amputation of the trial limb (above the knee, knee-ankle amputation, below the ankle amputation/toe amputation) | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
Change in Rutherford classification of the trial limb compared to baseline at first dose | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
  The Rutherford classification is a standardized system used to assess the severity of peripheral arterial disease (PAD) in the trial limb. It ranges from category 0 (asymptomatic) to category 6 (ischemic rest pain with gangrene). Higher categories indicate more severe disease. The change in Rutherford classification will be measured by comparing the classification at the first dose to the baseline classification.
Change in rest pain of the trial limb assessed by Numeric Rating Scale (NRS) compared to baseline at first dose | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose
  The NRS is a pain assessment tool that ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain. A higher score on the NRS indicates worse pain. The change in rest pain will be determined by comparing the NRS score at the first dose to the baseline NRS score.
Change in ulceration/necrosis of the trial limb compared to baseline at first dose | Every 3±1 months after enrollment, continuing until at least 36 months after the first dose

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - zhongshan Hospital Affiliated of Dalian University, Dalian, Shenyang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40221835/